CLINICAL TRIAL: NCT03282123
Title: An Open-Label, Multi-Site Phase 2 Study of the Safety and Effect of Manualized MDMA-Assisted Therapy for the Treatment of Severe Posttraumatic Stress Disorder
Brief Title: Open Label Multi-Site Study of Safety and Effects of MDMA-assisted Therapy for Treatment of PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-16
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Results first posted 2021-07-29 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: PTSD
Keywords: MDMA; methylenedioxymethamphetamine; therapy; midomafetamine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Three sessions of MDMA-assisted therapy with flexible dose of MDMA (80 to 120 mg with optional supplemental half-dose)
Masking Description: This study will be open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MDMA-assisted therapy (Experimental): Three sessions of MDMA-assisted therapy with flexible dose of midomafetamine HCl from 80 to 120 mg and optional supplemental dose half that of initial dose 1.5 to 2 hours later
  Interventions: Drug: Midomafetamine; Behavioral: Manualized therapy

INTERVENTIONS:
Drug: Midomafetamine — 80 to 120 mg MDMA
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA
Behavioral: Manualized therapy — Non-directive therapy conducted during MDMA-assisted therapy session

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted therapy is safe and effective in people diagnosed with at least severe PTSD.

The main question it aims to answer is: Do three open-label sessions of MDMA-assisted therapy reduce PTSD symptoms?

Participants will receive three non-drug preparatory sessions followed by three sessions of MDMA-assisted therapy. Each MDMA-assisted therapy session is followed by three non-drug integrative therapy sessions.

DETAILED DESCRIPTION:
This multi-site, open-label, Phase 2, lead-in study assesses the safety and efficacy of MDMA-assisted therapy in participants diagnosed with at least severe posttraumatic stress disorder (PTSD). Therapy teams that have been identified and trained to work on the sponsor's planned Phase 3 studies will treat at least one open-label participant in this study.

This study will compare the effects of three open-label manualized Experimental Sessions of psychotherapy assisted by flexible doses of MDMA. Initial doses per Experimental Session include 80 mg or 120 mg of MDMA compounded with lactose, followed 1.5 to 2 hours later by a supplemental half-dose (40 mg or 60 mg). Total amounts of MDMA to be administered per Experimental Session range from 80 mg to 180 mg. This ~12-week Treatment Period is preceded by three Preparatory Sessions. During the Treatment Period, each Experimental Session is followed by three Integrative Sessions of non-drug psychotherapy. The Primary Outcome measure is the change in Clinician Administered PTSD Scale for DSM 5 (CAPS-5) from Baseline to Primary Endpoint (Visit 19).

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old
* Are fluent in speaking and reading the predominantly used or recognized language of the study site
* Agree to have study visits recorded, including Experimental Sessions, Independent Rater assessments, and non-drug psychotherapy sessions
* Must provide a contact (relative, spouse, close friend or other caregiver) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.

Must agree to inform the investigators within 48 hours of any medical conditions and procedures

* If of childbearing potential, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 10 days after the last Experimental Session.
* Must not participate in any other interventional clinical trials during the duration of the study,
* Must be willing to remain overnight at the study site after each Experimental Session and be driven home after, and commit to medication dosing, therapy, and study procedures
* Meet DSM-5 Criteria for Severe PTSD

Exclusion Criteria:

* Are not able to give adequate informed consent
* Have uncontrolled hypertension
* Have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms] corrected by Bazett's formula)
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Have evidence or history of significant medical disorders
* Have symptomatic liver disease
* Have history of hyponatremia or hyperthermia
* Weigh less than 48 kilograms (kg)
* Are pregnant or nursing, or are of childbearing potential and are not practicing an effective means of birth control.
* Meet DSM-5 criteria for active substance use disorder for any substance other than caffeine or nicotine
* Have used Ecstasy (material represented as containing MDMA) more than 10 times within the last 10 years or at least once within 6 months of the first Experimental Session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Mithoefer, MD, Study Director — MAPS Public Benefit Corp.
Locations (12):
- United States (12):
  - New School Research LLC, North Hollywood, California
  - San Francisco Insight and Integration Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Aguazul-Blue Water Inc., Boulder, Colorado
  - Wholeness Center, Fort Collins, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Ray Worthy Psychiatry LLC, New Orleans, Louisiana
  - Trauma Research Foundation, Brookline, Massachusetts
  - New York University, New York, New York
  - Affective Care, New York, New York
  - Zen Therapeutic Solutions, LLC, Mt. Pleasant, South Carolina
  - University of Wisconsin at Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christie D, Yazar-Klosinski B, Nosova E, Kryskow P, Siu W, Lessor D, Argento E. MDMA-assisted therapy is associated with a reduction in chronic pain among people with post-traumatic stress disorder. Front Psychiatry. 2022 Nov 3;13:939302. doi: 10.3389/fpsyt.2022.939302. eCollection 2022. PMID 36405923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through print and internet advertisements, referrals from other psychiatrists, psychotherapists, or physicians, and by word of mouth. The sponsor monitored demographics on an ongoing basis and encouraged diversity in enrollment by communicating with sites
Groups:
- MDMA-assisted Psychotherapy: Three sessions of MDMA-assisted psychotherapy with flexible dose of MDMA from 80 to 120 mg and optional supplemental dose half that of initial dose 1.5 to 2 hours later
  MDMA: 80 to 120 mg MDMA
  Psychotherapy: Non-directive psychotherapy conducted during MDMA-assisted psychotherapy session
Period: Overall Study
Arm/Group | MDMA-assisted Psychotherapy
Started | 38
Completed | 33
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: Safety Set
Arm/Group | MDMA-assisted Psychotherapy
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.42 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 24
  More than one race | 2
  Unknown or Not Reported | 0
Baseline CAPS-5 Total Severity Score [Mean (Standard Deviation); unit: score on a scale] | 45.4 (6.70)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Visit 19 in CAPS-5 Total Severity Scores
Description: The Clinician-Administered PTSD Scale for DSM-V (CAPS-5) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-5. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Baseline to 18 weeks post-enrollment
Population: Safety Set
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- MDMA-assisted Therapy: Three sessions of MDMA-assisted therapy with flexible dose of MDMA from 80 to 120 mg and optional supplemental dose half that of initial dose 1.5 to 2 hours later
  MDMA: 80 to 120 mg MDMA
  Psychotherapy: Non-directive therapy conducted during MDMA-assisted therapy session
Arm/Group | MDMA-assisted Therapy
Number analyzed (Participants) | 33
score on a scale | -30.49 [-34.16 to -26.83]

2. Secondary Outcome: Change From Baseline to Visit 19 in Adapted SDS Total Score
Description: The Sheehan Disability Scale (SDS) is a clinician-rated assessment of functional impairment that was adapted for the purposes of this study to limit missing item-level data as per the FDA requirements and included use of the three-item mean as the total score and imputation of work-related impairment. The SDS is a 3-item scale measuring the severity of disability in the domains of work, family life/home responsibilities and social/leisure activities, with each item scored on a ten-point Likert scale from 0 ('not at all impaired') to 10 ('very severely impaired'). The SDS total score was the mean of the 3 item responses. The SDS total score ranged from 0 to 10, with higher scores indicating greater functional impairment.
Time Frame: Baseline to 18 weeks post-enrollment
Population: Safety Set
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- MDMA-assisted Psychotherapy: Three sessions of MDMA-assisted therapy with flexible dose of MDMA from 80 to 120 mg and optional supplemental dose half that of initial dose 1.5 to 2 hours later
  MDMA: 80 to 120 mg MDMA
  Psychotherapy: Non-directive therapy conducted during MDMA-assisted therapy session
Arm/Group | MDMA-assisted Psychotherapy
Number analyzed (Participants) | 33
score on a scale | -4.88 [-5.7 to -4.06]

ADVERSE EVENTS:
Time Frame: All treatment-emergent adverse events until end of study (approximately 5 months)
Arm/Group | MDMA-assisted Psychotherapy
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 1/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDMA-assisted Psychotherapy (N=33)
Suicide attempt (Psychiatric disorders) | 1 (1) — One participant with a history of suicidal ideation and two unsuccessful suicide attempts prior to the study attempted suicide 28 days after the third experimental session.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MDMA-assisted Psychotherapy (N=33)
Palpitations (Cardiac disorders) | 3
Vision Blurred (Eye disorders) | 2
Abdominal Discomfort (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 11
Dry Mouth (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 8
Temperature Intolerance (General disorders) | 2
Chest Discomfort (General disorders) | 2
Pain (General disorders) | 2
Decreased Appetite (Metabolism and nutrition disorders) | 4
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 18
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 3
Nystagmus (Nervous system disorders) | 8
Headache (Nervous system disorders) | 22
Dizziness (Nervous system disorders) | 5
Paraesthesia (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 11
Restlessness (Psychiatric disorders) | 3
Panic Reaction (Psychiatric disorders) | 2
Flashback (Psychiatric disorders) | 3
Bruxism (Psychiatric disorders) | 3
Suicidal Ideation (Psychiatric disorders) | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 3
Viral upper respiratory tract infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Chills (General disorders) | 2
Pyrexia (General disorders) | 2
Nasopharyngitis (Infections and infestations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Taste disorder (Nervous system disorders) | 2
Micturition urgency (Renal and urinary disorders) | 2
Visual impairment (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT03282123/Prot_003.pdf
  • Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT03282123/SAP_001.pdf
  • Informed Consent Form (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT03282123/ICF_004.pdf